CLINICAL TRIAL: NCT05430113
Title: Spinal Cord Stimulation for the Treatment of Motor Deficits in People With Spinal Muscular Atrophy
Brief Title: Spinal Cord Stimulation in Spinal Muscular Atrophy
Acronym: SCSinSMA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marco Capogrosso (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor-Investigator, Marco Capogrosso, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY21080158
Record Dates: First submitted 2022-04-12; First posted 2022-06-24 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Spinal Muscular Atrophy Type 3; Spinal Muscular Atrophy Type 4
Keywords: Spinal Muscular Atrophy; Spinal Cord Stimulation
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label study performed to quantify variables that are predictive of the efficacy of spinal cord stimulation to improve motor control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Spinal Cord Stimulation (Experimental): All patients will receive FDA-approved percutaneous spinal cord stimulation leads implanted in the epidural (T12-L2 vertebra) space. The leads will be connected to external stimulators (either FDA-approved or human-grade research stimulator with safety features) during research activities.
  Interventions: Device: Spinal Cord Stimulator (octopolar Medtronic Vectris Leads)

INTERVENTIONS:
Device: Spinal Cord Stimulator (octopolar Medtronic Vectris Leads) — 2-4 leads FDA-approved for treatment of symptoms of refractory pain

SUMMARY:
Spinal cord stimulation (SCS) has shown remarkable efficacy in restoring motor function in people with spinal cord injury by recruiting afferent input to enhance the responsiveness of spared neural circuits to residual cortical inputs. This pilot will test if SCS can show evidence to improve motor deficits in people with type 3 or 4 spinal muscular atrophy (SMA). The investigators will enroll up to six subjects with Type 3 or 4 SMA aged 16 or older that show quantifiable motor deficits of the legs but are able to stand independently. The investigators will then implant the subjects with percutaneous, bilateral, linear spinal leads near the lumbar spinal cord for a period of up to 29 days. Although these leads are not optimized for motor function but rather for their clinically approved indication of treating pain, the investigators believe they provide a safe technology enabling our team to perform scientific measurement necessary to evaluate potential for effects of SCS in motor paralysis with SMA. After the end of the study, the leads will be explanted.

DETAILED DESCRIPTION:
The investigators plan to 1. verify that spinal cord stimulation increases hip muscle strength in subjects with SMA, 2. verify that spinal cord stimulation improves motor control in subjects with SMA, 3. verify that spinal cord stimulation induces measurable changes in spinal circuits and motoneuron recruitment properties in the 29 day course of implantation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject or subject's parent or legal guardian (for minor subjects) has provided written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization, where applicable, prior to any study-related procedures. Minor subjects will be asked to give written assent according to local requirements.
2. Subject has a diagnosis of 5q-autosomal recessive SMA confirmed by determination of a genetic deletion in the SMN1 gene (5q12.2-q13.3)
3. Subject is diagnosed as having Type 3 or Type 4 SMA based on the following criteria

   1. Disease manifested after 18 months of age
   2. Disease manifested after ambulation was acquired
4. Subject is ≥16 years of age and < 65 years of age
5. Subject is able to stand independently for ≥3 seconds
6. RHS score lower or equal to 65
7. Subject (and subject's parent or legal guardian if subject is a minor) is willing and able to comply with scheduled visits and study procedures

Exclusion Criteria:

1. Subject has deformation of the spinal canal preventing lead implantation as judged by the study neurosurgeon
2. Subject has size of spinal canal that is insufficient for lead implantation as judged by the study neurosurgeon
3. Subject has moderate or severe joint contractures that would affect ability to perform study measures
4. Subject has severe behavioral or cognitive problems that preclude participation in the study, in the opinion of the investigator
5. Subject has previous or ongoing medical condition, medical history, physical findings or laboratory abnormalities that could affect safety of anesthesia or the procedures, make it unlikely that intervention or follow-up will be correctly completed or impair the assessment of study results, in the opinion of the investigator
6. Female subjects are pregnant or breastfeeding
7. Subject has severe claustrophobia
8. Subject is on anticoagulant, anti-spasticity or anti-seizure medication within 4 weeks of lead implantation or requires these medications during the treatment phase of the study
9. Subject has medical implant that precludes magnetic resonance imaging

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Muscle Weakness | 29 days
  Isometric torque: measure the isometric torque produced by the subject at the hip during hip-flexion. Comparison of SCS-on with SCS-off performance. Success Criteria: ≥20% increased torque production over SCS-off baseline as measured during single-joint isometric torque.
Number and Severity of Adverse Events | 29 days
  Success Criteria: no serious adverse event related to the stimulation or intolerable adverse event reported

SECONDARY OUTCOMES:
Muscle Weakness 2 | 29 days
  Muscle activation: measure surface EMGs produced by the subjects during isometric movements of the hip, knee, and ankle in the HUMAC Norm and compare SCS-on with SCS-off performances. Meaningful Change:<20% EMG RMS compared to SCS-on.
Motor Function ROM | 29 days
  Range of Motion (ROM): Meaningful Change: increase of >20% of the hip joint (if available) and the knee joint (if available) during SCS against SCS-off as measured by the HUMAC NORM during single-joint isotonic trials.
Motor Function: 6-Minute Walk Teset | 29 days
  6 minute walk test: perform the 6-minute walk test with SCS-on and SCS-off and distance between SCS-on and SCS-off is set to 24 m. If not ambulator, any increased ambulation distance from SCS-off condition.
Motor Function RHS | 29 days
  The Revised Hammersmith Functional Scale is a further refined version of the Hammersmith Functional Motor Scale Extended and includes specific items focused on lower-limb motor control such as hip-flexion, standing and walking a that are particularly relevant for the type III population of study. The scale is a 36 item performance evaluation, with a score range from 0-69 in which higher scores indicate better performance.
  Meaningful Change: ≥2 point improvement. Compare outcomes between SCS-on and SCS-off. Motor Function Measure 32. The 32 items MFM is often used in trials of neuromuscular disorders, hence it provides a meaningful comparison against outcomes of other trials. Meaningful Change: ≥2 point improvement. Compare outcomes between SCS-on and SCS-off.
Motor Function: Fatigue | 29 days
  Fatigue will be assessed during motor function tests.
Discomfort/Pain | 29 days
  Patients will be asked to provide a score from 1 to 10 where a greater number indicates a greater amount of discomfort for each stimulation configuration. Spinal cord stimulation produces tingling sensations and other type of sensory phenomena. It is important to document that stimulation intensities required to improve motor function remain within a range of non-painful sensations.
Sensorimotor Network Structure Density | 29 days
  The investigators will perform High-definition Diffusion Weighted Imaging to quantify Fractional Anisotropy as a measurement of axon density in the brain and spinal cord pre and post study.
Impression | 29 days
  The investigators will collect subjects and therapist feedback on how the technology is performing and what they would want to modify using The Clinical Global Impression Scale, a scale of 1-7 where a lower number indicates better performance and a higher number indicates more greatly impacted by their disease.
Sensorimotor Network Structure Integrity | 29 days
  The investigators will perform High-definition Diffusion Weighted Imaging to quantify Fractional Anisotropy as a measurement of axon integrity in the brain and spinal cord pre and post study.
Sensorimotor Network Function | 29 days
  The investigators will perform resting state and motor-task functional MRI of the brain and spinal cord to quantify neural network activation at rest and during the execution of simple motor task such as leg muscle contraction.
Cortico-spinal Tract Integrity | 29 days
  The investigators will measure muscle evoked potential consequent to Transcranial Magnetic Stimulation of the cortico-spinal tract to assess integrity of the cortico-spinal tract.
Spinal Circuit Excitability | 29 days
  The investigators will measure H-reflexes of leg muscles to quantify excitability of spinal motoneurons to stimulation of primary sensory afferents pre and post-study. Expected Result: Our main scientific hypothesis is that SCS will restore monosynaptic responses of weak spinal motoneurons, thus increasing H-reflex responses pre and post-study.
Motoneuron Firing Rates | 29 days
  The investigators will use high-density EMGs on leg muscles to calculate firing rates of single spinal motoneuron discharge during isometric maximal voluntary contractions.
Motor Firing Number | 29 days
  The investigators will use high-density EMGs on leg muscles to calculate the number of firing rates of single spinal motoneuron discharge during isometric maximal voluntary contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Capogrosso, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available at the end of the trial upon publication of the first manuscript. Estimation is 2 years from enrollment of first participant
Access Criteria: Data must be directly requested to the PI and will be shared upon completion of necessary data sharing agreement to protect confidential patient information

REFERENCES:
- [Derived] Prat-Ortega G, Ensel S, Donadio S, Borda L, Boos A, Yadav P, Verma N, Ho J, Carranza E, Frazier-Kim S, Fields DP, Fisher LE, Weber DJ, Balzer J, Duong T, Weinstein SD, Eliasson MJL, Montes J, Chen KS, Clemens PR, Gerszten P, Mentis GZ, Pirondini E, Friedlander RM, Capogrosso M. First-in-human study of epidural spinal cord stimulation in individuals with spinal muscular atrophy. Nat Med. 2025 Apr;31(4):1246-1256. doi: 10.1038/s41591-024-03484-8. Epub 2025 Feb 5. PMID 39910271